CLINICAL TRIAL: NCT00058981
Title: Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Investigate the Safety and Tolerability as Well as the Immunological and Clinical Efficacy of Multiple Subcutaneous Doses of DiaPep277 in LADA Subjects
Brief Title: Safety, Tolerability, Immunological and Clinical Efficacy of Multiple Subcutaneous Doses of DiaPep277 in Latent Autoimmune Diabetes in Adults (LADA)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: DeveloGen Israel, Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 702/PO
Record Dates: First submitted 2003-04-15; First posted 2003-04-24 (Estimated); Last update posted 2009-03-19 (Estimated); Status verified 2009-03

CONDITIONS: Diabetes, Autoimmune
Keywords: Diabetes; LADA; latent autoimmune diabetes in adults
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Latent Autoimmune Diabetes in Adults

INTERVENTIONS:
Drug: DiaPep277

SUMMARY:
Randomized, double-blind, parallel-group study to evaluate safety and efficacy of multiple subcutaneous doses of DiaPep277 in patients with Latent Autoimmune Diabetes in Adults (LADA). Study medication will be administered at time 0, 1 and 3 months, and then every 3 months for a total of 8 administrations. The total duration of the trial is 24 months (treatment for 18 months and follow-up for an additional 6 months). Patients will be male or female between the ages of 30 and 65 years, inclusive, within 2 to 60 months of the diagnosis of diabetes mellitus. Subjects must be positive for glutamic acid decarboxylate (GAD) autoantibodies. At the Screen Visit (Visit 2), all subjects will be asked to discontinue their use of all oral antidiabetic medications with the exception of metformin. The subjects will be placed on a stable regimen of insulin and diet (plus metformin if needed). Prior to the Baseline Visit (Visit 3), diabetic control must be achieved by diet and insulin (plus metformin if needed).

ELIGIBILITY:
Inclusion Criteria

Subjects meeting all of the following inclusion criteria at screening should be considered for admission to the study:

* The subject has a diagnosis of diabetes mellitus according to WHO classification for more than 2 months and less than 5 years before enrollment.
* The subject's diabetes has been controlled by diet and insulin (plus metformin if needed) for 2 or more weeks (14 days) prior to the Baseline Visit (Visit 3).
* The subject is a male or female aged 30 to 65 years. If female and not postmenopausal, the subject is not pregnant and will use effective contraceptive methods throughout the study.
* The subject is positive for GAD autoantibodies, defined as a level greater than the 99th percentile of the GAD antibody index of a normal control population for the laboratory (e.g., GAD antibody index equal to 0.085).
* The subject has a fasting C-peptide level 0.30 nmol/L or greater or 0.9 ng/mL at the time of the Screen Visit (Visit 1 or 2).

Exclusion Criteria

Subjects meeting any of the following exclusion criteria at screening will not be enrolled in the study:

* The subject has any significant diseases or conditions, including psychiatric disorders and substance abuse that, in the opinion of the site investigator, are likely to affect the subject's response to treatment or their ability to complete the study.
* The subject has a history of any kind of malignant tumor.
* The subject has secondary diabetes mellitus.
* Within 2 weeks or 14 days of the Baseline Visit or during randomized treatment, the subject takes an oral anti-diabetic medication other than metformin to treat his/her diabetes.
* The subject has clinical evidence of any diabetes-related complication that in the opinion of the site investigator would interfere with the subject's participation in and/or completion of the study.
* The subject has a history of allergy or asthma that in the opinion of the site investigator would interfere with the subject's participation in and completion of the study.
* The subject has a known immune deficiency from any disease, or a condition associated with an immune deficiency.
* The subject is receiving immunosuppressive or immunomodulating agents or cytotoxic therapy, or any medication that, in the opinion of the site investigator, might interfere with the study.
* The subject is a pregnant woman or a woman who is planning to become pregnant.
* The subject has any of the following:

  * chronic hepatitis or liver cirrhosis, or any other chronic liver disease
  * is known to test positive for hepatitis B antigens or hepatitis C antibodies
  * has abnormal liver function, defined as serum AST or ALT 3 times or more the upper limit of normal
* The subject is a known or suspected drug abuser.
* The subject has influenza-like symptoms on the day of dosing.
* The subject is known to test positive for HIV antibodies.
* The subject has chronic hematologic disease.
* The subject has impaired renal function (serum creatinine greater than 1.4 mg/dL).
* The subject has severe ketonuria (+++ on urine stix testing; ++ on repeated urine stix testing).
* The subject has a BMI greater than 40kg/m2.
* The subject has hyperlipidemia (fasting serum triglycerides >1000 mg/dL). Suitable medical therapy for treatment of hyperlipidemia is allowed.
* The subject has received any investigational drug within 3 months prior to Visit 1.
* The subject has had a severe blood loss (400 mL or more, e.g., blood donation) within 2 months before the first dosing of the study medication.
* The subject is a breast-feeding mother or planning to breast-feed.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2002-10; Primary Completion 2007-03 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry P Palmer, MD, Principal Investigator — University of Washington; Dana Elias, PhD, Study Director — DeveloGen Israel, Ltd.
Locations (7):
- United States (7):
  - University of Alabama at Birmingham Endocrinology Department, Birmingham, Alabama
  - University of Colorado Hospital Endocrinology Practice, Aurora, Colorado
  - University of Kentucky Department of Internal Medicine, Lexington, Kentucky
  - Washington University School of Medicine Endocrinology/Metabolic Dept, St Louis, Missouri
  - North Shore Diabetes and Endocrine Associates, New Hyde Park, New York
  - Diabetes & Glandular Disease Research Associates, San Antonio, Texas
  - DVA Puget Sound Health Care System Endocrinology (III) Department, Seattle, Washington

REFERENCES:
- [Derived] Pozzilli P, Raz I, Peled D, Elias D, Avron A, Tamir M, Eren R, Dagan S, Cohen IR. Evaluation of long-term treatment effect in a type 1 diabetes intervention trial: differences after stimulation with glucagon or a mixed meal. Diabetes Care. 2014;37(5):1384-91. doi: 10.2337/dc13-1392. Epub 2014 Jan 9. PMID 24408401 (Retraction: PMID 25538318 Diabetes Care. 2015 Jan;38(1):179)